CLINICAL TRIAL: NCT01941303
Title: Radical Re-irradiation of Recurrent NSCLC - Analysis of Outcome and Toxicity.
Brief Title: Analysis of Treatment Outcome and Toxicity in Non-small Cell Lung Cancer Patients Wither-irradiated to a High Dose for Recurrent Disease
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Irradiation treatment outcome; NCT01930825 (obsolete NCT alias)
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced stage non-small cell lung cancer patients

SUMMARY:
As one of the few centers, MAASTRO also aggressively re-treats patients with recurrent non-small cell lung cancer. Even after primary radical treatment to high doses, re-irradiation (with concurrent chemotherapy) is also given in curative intent, thus again using high doses of radiation.

Publications on high-dose re-irradiation of lung cancer patients are scarce, and outcome and toxicity for patients treated in MAASTRO are unknown at present. This study will provide knowledge on benefit and risks of such a therapeutic approach.

DETAILED DESCRIPTION:
MAASTRO clinic is a leader in the (individual) management of patients with lung cancer. This has resulted in major publications in the past on individualized (chemo)radiotherapy for (NSCLC) [van Baardwijk 2006 and 2010]. As one of the few centers, MAASTRO also aggressively re-treats patients with recurrent non-small cell lung cancer. Even after primary radical treatment to high doses, re-irradiation is also given in curative intent, thus again using high doses of radiation.

Publications on this topic are rare. Most reports address the results of palliative re-irradiation of NSCLC [Ebara 2007, Jackson 1987, Montebello 1993, Tada 2005]. The ones available on re-irradiation with curative intent used outdated techniques [Okamoto 2002, Wu 2003]. Only one recent publication has analyzed the results of 37 NSCLC patients of whom 9 were re-irradiated with at least 50 Gy using helical tomotherapy [Kruser in press].

The results of radical re-irradiation applying highly conformal radiation techniques within MAASTRO are unknown. This study will provide knowledge on benefit and risks of such a therapeutic approach. Furthermore, it may provide enough evidence to initiate a Phase II/III clinical trial for re-irradiation of NSCLC patients with curative intent.

ELIGIBILITY:
Patients with advanced stage non-small cell lung cancer treated to higher doses of irradiation (i.e. EQD2>50Gy) twice: in the primary and recurrent setting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-small cell lung cancer undergoing chest irradiation (with chemotherapy) to a radical dose twice: in the primary and the recurrent setting.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year after radiotherapy
  Measuring survival by checking if patients are alive.
Locoregional control | 1 year after radiotherapy
  Measuring locoregional control by checking pt for progression
Progression-free survival | 1 year after radiotherapy
  Checking patients for progression

SECONDARY OUTCOMES:
Pulmonary toxicity | 1 year after radiotherapy
  Checking patients for pulmonary adverse events
Oesophageal toxicity | 1 year after radiotherapy
  Checking patients for oesophageal adverse events
Other dose-limiting or burdensome toxicity | 1 year after radiotherapy
  Checking patients fortoxicity which causes problems with regard to radiotherapy-dose or is otherwise burdensome

CONTACTS AND LOCATIONS:
Overall Officials: Esther Troost, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands